CLINICAL TRIAL: NCT00856063
Title: Feasibility and Utility of Autonomic Correlates of Impulsivity in Preschool Children With Attention Deficit Hyperactivity Disorder (ADHD): Extending Translational Research Skills
Brief Title: Autonomic Correlates of Impulsivity for Preschool Children With Attention Deficit Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: ACTREC JG - 08
Record Dates: First submitted 2009-03-03; First posted 2009-03-05 (Estimated); Last update posted 2012-07-09 (Estimated); Status verified 2012-07

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Attention Deficit Hyperactivity Disorder; Atomoxetine; Electrodermal Response; Impulsivity; Preschool Children
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Impulsive Behavior | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: atomoxetine (or placebo) — Each child will be randomized to receive either ATMX or placebo in the 1st crossover phase followed by the alternative drug condition in the 2nd crossover phase. The study drug (ATMX or placebo) will be administered BID and will be titrated blindly based on clinical response and tolerability. ATMX will be initiated at 0.5 mg/kg/day for 3 days. Based on clinical response, ATMX dose will be titrated to 0.8 mg/kg/day during week 1, 1.4 mg/kg/day during week 2, and a maximum of 1.8 mg/kg/day during week 3, unless serious untoward effects intervene.

SUMMARY:
The goal of this pilot feasibility and utility study is to develop and validate a method that is reproducible over time for assessing biobehavioral and autonomic markers of impulsivity and their utility in assessing treatment outcome in preschool children with ADHD.

DETAILED DESCRIPTION:
Assessing biological markers of ADHD among preschoolers has the potential to elucidate biology-environment interactions, which may have important implications for treatment, and for our understanding of the etiology of ADHD. Although impulsivity is highly heritable, long-term changes in biological systems implicated in impulsive behavior can be effected through intervention as shown by a 61% increase in electrodermal activity 6-8 years later in at-risk preschool children who were randomized to the intervention condition compared with controls randomized to no treatment condition. Early intervention may therefore be essential if dysregulated trajectories in responding within these systems are to be prevented and/or altered.

Atomoxetine (ATMX) blocks the NE transporter (NET), and increases extracellular levels of NE throughout the brain. It is the first nonstimulant drug approved by the FDA for the treatment of ADHD. Recent clinical studies have shown that ATMX significantly reduces symptoms of ADHD as observed by parents and teachers. ATMX has been shown to improve response inhibition in ADHD.

In the proposed research, pre- and post-treatment bio-behavioral and autonomic markers of impulsivity will be assessed in preschool children with ADHD who participate in a double blind, randomized, placebo-controlled crossover treatment with a selective NET inhibitor, atomoxetine, and placebo.

ELIGIBILITY:
Inclusion Criteria:

* 48-70 month old children.
* diagnosis of ADHD based on caregiver interview and confirmed by clinical interview.
* level of hyperactivity/impulsivity at home and school (if relevant)
* significant impairment in everyday functioning.

Exclusion Criteria:

* prior failed treatment with an adequate trial of atomoxetine (ATMX)or known hypersensitivity to ATMX.
* contraindication to ATMX.
* comorbid psychiatric diagnoses of mental retardation,pervasive developmental disorders, bipolar disorder, major depressive disorder, panic disorder, obsessive compulsive disorder, post traumatic stress disorder, psychotic disorder, or suicidality.
* concurrent treatment with other medications that have central nervous system effects or that affect performance, e.g., antidepressants, antipsychotics, alpha-agonists, adrenergic blockers, decongestant or sympathomimetics, sedating antihistamines, or lithium carbonate.
* taking monoamine oxidase inhibitors (MAOI) or less than 2 weeks have passed since MAOI treatment was discontinued.
* medical condition which may interfere with involvement with the study or would be affected negatively by ATMX, including narrow angle glaucoma, significant hepatic or cardiac disease,high heart rate and blood pressure.
* current history of physical, sexual, or emotional abuse.
* has taken an investigational drug within the last 30 days.

Ages: 48 Months to 70 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2009-03; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Hyperactive-Impulsive subscale of SNAP-IV (Swanson, Nolan and Pelham [SNAP] Questionnaire) | 3-4.5 months

SECONDARY OUTCOMES:
Children's Global Assessment Scale (C-GAS) | 3-4.5 months
Electrodermal response (EDR) | 3-4.5 months
Response inhibition task | 3-4.5 months

CONTACTS AND LOCATIONS:
Overall Officials: Jaswinder Ghuman, M.D., Principal Investigator — University of Arizona